CLINICAL TRIAL: NCT01732601
Title: Intensive Outpatient Protocol for High Risk Suicidal Teens
Brief Title: Intensive Outpatient Services for Teens
Acronym: INVEST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Anthony Spirito, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01MH097703-01 (NIH); 1R01MH097703-01 (NIH)
Record Dates: First submitted 2012-11-13; First posted 2012-11-26 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Depression; Suicide
Keywords: Suicide Attempt; Suicidal Ideation; NSSI; Substance Use
MeSH Terms: conditions — Depression; Suicide; Suicide, Attempted; Suicidal Ideation; Substance-Related Disorders | interventions — Standard of Care; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive Outpatient CBT (Experimental): Intensive CBT for both parents and adolescents as well as family sessions to increase communication.
  Interventions: Behavioral: Intensive Outpatient CBT
- Standard Care (Active Comparator): Standard Treatment in the Community
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Intensive Outpatient CBT — Sessions will be delivered 1-2 times a week for the first 4-6 weeks, based on need, and then weekly until 6 months. Therapy can continue up until one year.
  Other Names: Intensive CBT for High Risk Teens with a mood disorder
  Arms: Intensive Outpatient CBT
Behavioral: Standard Care — Treatment at step-down facilities
  Other Names: Treatment as Usual
  Arms: Standard Care

SUMMARY:
This study will identify the effectiveness of an intensive treatment program for teens who are at high risk for harming themselves.

DETAILED DESCRIPTION:
Suicidal ideation and behavior are the primary reasons for emergency psychiatric care and inpatient psychiatric hospitalization in this country. These expensive contacts with the health care system effectively address acute suicidality for many adolescents but there is a significant subset of suicidal patients that have continued suicidality. This study will target teens that are at risk for re-hospitalization based on continued suicidal ideation, their mood and another risk factor such as self-harm or substance use. These risk factors have been shown to increase risk for continued suicidal behavior and expensive contacts with the health care system. This protocol has been designed to determine whether Intensive Cognitive Behavioral Therapy (CBT), which was designed to treat adolescents with a mood disorder, suicidal ideation, and substance use, will result in better treatment outcomes compared to standard care in the community. The Intensive CBT condition will be delivered by a team of two licensed mental health therapists over the course of one year and will work with both the teen and parent. The standard care condition will receive treatment in the community. One hundred-and fifty adolescents (38 a year) will be recruited from several inpatient and partial hospital locations. Each adolescent will receive a thorough baseline assessment to determine whether they are appropriate for the study and will be assigned to either the Intensive CBT condition or treatment within the community. Both groups of teens will receive follow-up assessments at 6, 12, and 18 months to identify how they are doing over time.

ELIGIBILITY:
Inclusion Criteria:

* Current Mood Disorder and suicidal ideation and one of the following
* NSSI
* Suicide Attempt
* Substance Use

Exclusion Criteria:

* Intelligence Quotient < 80
* Diagnosis of psychotic disorder, pervasive developmental disorder, obsessive-compulsive disorder, bulimia nervosa or anorexia nervosa
* Adolescent use of illicit "hard" substances such as cocaine, heroine, and opiates 13 or more times over the prior 90 days

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Suicide attempts | Measured at 18 months from Baseline
  Self-report by parents or teens of a suicide attempt occurring in the follow-up period

SECONDARY OUTCOMES:
Depressed mood as assessed by the Children's Depression Rating Scale - Revised | Measured at 18 months from Baseline
  Depressed mood as determined by clinical interview

OTHER OUTCOMES:
Other self harm behaviors including Nonsuicidal self-injury (NSSI) substance abuse | Measures 18 months from Baseline
  Self report of behaviors considered self-harming including self-inflicted behaviors such as cutting with no suicidal intent or excessive substance use with negative consequences to the individual

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Spirito, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Esposito-Smythers C, Wolff JC, Liu RT, Hunt JI, Adams L, Kim K, Frazier EA, Yen S, Dickstein DP, Spirito A. Family-focused cognitive behavioral treatment for depressed adolescents in suicidal crisis with co-occurring risk factors: a randomized trial. J Child Psychol Psychiatry. 2019 Oct;60(10):1133-1141. doi: 10.1111/jcpp.13095. Epub 2019 Jul 21. PMID 31328281